CLINICAL TRIAL: NCT05767775
Title: Synovial and Adipose Tissue Derived Biomarkers of Clinical Response in Overweight/Obese Patients With Active Rheumatoid Arthritis Under JAK/STAT Inhibition
Brief Title: Synovial and Adipose Tissue Composition in Overweight/Obese Patients With Active Rheumatoid Arthritis Under JAK/STAT Inhibition
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Alivernini Stefano, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2237
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: synovial tissue; adipose tissue; JAK-inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients with BMI≥ 25 eligible to Tofacitinib
  Interventions: Other: Assessment of synovial- and adipose tissue-derived inflammatory biomarkers
- RA patients with BMI<25 eligible to Tofacitinib
  Interventions: Other: Assessment of synovial- and adipose tissue-derived inflammatory biomarkers

INTERVENTIONS:
Other: Assessment of synovial- and adipose tissue-derived inflammatory biomarkers — Parafﬁn-embedded synovial tissue (ST) specimens will be stained for H&E and other sections will be stained for CD68, CD21, CD20, CD3, CD31 and Masson Trichrome Goldner with light green to assess the microanatomical organization of resident synovial inflammatory cells. Some synovial samples will be used for tissue resident macrophages subpopulations analysis using FACS gated on their expression of the CD64+/CD11b+/MHC-ClassII+/CD206+/-/Lineage-.
  Each RA patient reaching a stable clinical (DAS<1.6 for at least two different evaluations 6 months apart) and imaging (PDUS negative signal) remission under Tofacitinib treatment will undergo synovial biopsy and each synovial tissue sample will be processed as above.
  Plasma levels of adipokines will be tested through ELISA method at baseline, 3, 6 and 12 months of follow-up in all patients.

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic autoimmune disease that affects nearly 1% of the general population worldwide leading to joint inflammation, disability and increate mortality. Several factors are associated with disease activity and treatment outcomes. Among them, overweight/obesity status was demonstrated to be associated with higher risk of RA development and most importantly to different treatment response to biological DMARDs. Moreover, overweight/obese RA patients do show higher degree of synovial inflammation compared to lean RA patients. In this context, adipose tissue accumulation is associated with higher inflammatory burden through the secretion by activated mature adipocytes of adipokines with pro-inflammatory properties on innate and adaptive immune cells. Among them, Leptin is an important adipokine, released by mature adipocytes with multiple activating properties on immune cells as monocytes, macrophages, dendritic cells, T and B lymphocytes acting through the activation of its receptor LEPR via JAK/STAT pathway. In particular, leptin exerts its effects on macrophages populations through the promotion of M1 differentiation with pro-inflammatory phenotype. In our research hypothesis we expect that leptin levels does correlate with immunohistochemical scores of synovial inflammatory cells (CD68+, CD21+, CD20+ and CD3+) and CD31+ synovial vessels. Moreover, we expect that the inhibition of JAK/STAT signal using Tofacitinib may interfere with leptin activation action on resident synovial inflammatory cells expressing LEPR (as CD68+, CD20+ and CD3+) in particular restoring the M1/M2 phenotype ratio within resident macrophages populations. Finally, we expect that the inhibition of JAK/STAT signaling pathway by Tofacitinib will result in a significant reduction of synovitis degree in patients with higher leptin expression due to adipose tissue activation.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling 2010 ACR/EULAR classification criteria for Rheumatoid Arthritis.
* Patients with inadequate response to Methotrexate at the maximum tolerated dose (10-25 mg/week), or first bDMARD with at least moderate disease activity (DAS28>3.2), with disease duration <12 months or naïve to prior biologic therapy.
* Patients eligible to Tofacitinib according to the treating physician judgement.
* Stable low doses of prednisone (<5 mg/daily) since at least three months if necessary are allowed at the time of enrollment.

Exclusion Criteria:

* Severe and uncontrolled infections such as sepsis and opportunistic infections.
* Patients who are currently included in any interventional clinical trial in RA.
* RA patients treated with more than one biologics.
* Subjects who are impaired, incapacitated, or incapable of completing study-related assessments
* Subjects with active vasculitis of a major organ system, with the exception of rheumatoid nodules.
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, whether or not related to RA and which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
* Female subjects who have had a breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory, or other diagnostic evaluations.
* Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ. Existing non-melanoma skin cell cancers should be removed, the lesion site healed, and residual cancer ruled out before administration of the study drug.
* Subjects who currently abuse drugs or alcohol.
* Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
* Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
* Subjects who have received any live vaccines within 3 months of the anticipated first dose of study medication.
* Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis).
* Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be subjects with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with RA with inadequate response to Methotrexate at the maximum tolerated dose (10-25 mg/week), or first bDMARD with at least moderate disease activity (DAS28>3.2), with disease duration <12 months or naïve to prior biologic therapy. RA patients eligible to Tofacitinib according to the treating physician judgement. RA patients under stable low doses of prednisone (<5 mg/daily) since at least three months if necessary are allowed at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
DAS-remission achievement under Tofacitinib | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Rheumatology, Rome, Italy

IPD SHARING:
Plan to Share IPD: No